CLINICAL TRIAL: NCT03105375
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of X842 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of X842 in Human: A Single/Multiple Ascending Dose Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CX842A2101
Record Dates: First submitted 2017-03-01; First posted 2017-04-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
Keywords: Potassium competitive acid blocker; X842; Gastroesophageal reflux disease; Esophagitis; Intragastric pH; Acid inhibition
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: SAD and MAD study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single ascending dose of X842 (Experimental): Single ascending oral dose of X842 administered to subjects in cohorts. Cohorts are administered in sequence.
  Interventions: Drug: Single ascending dose of X842
- Multiple ascending dose of X842 (Experimental): Multiple ascending oral dose of X842 administered to subjects in cohorts. Cohorts are administered in sequence.
  Interventions: Drug: Multiple ascending dose of X842
- Losec (Active Comparator): Standard oral dose of omeprazole administered to subjects in one cohort.
  Interventions: Drug: Losec

INTERVENTIONS:
Drug: Single ascending dose of X842 — Each subject in a the same cohort will be assigned to the same single dose of X842. The subjects in the subsequent cohort will be assigned to a single dose of X842 based on safety and efficacy data generated from the previous cohort.
  Other Names: X842
  Arms: Single ascending dose of X842
Drug: Multiple ascending dose of X842 — Each subject in a the same cohort will be assigned to the same dose of X842 once daily for five days. The subjects in the subsequent cohort will be assigned to same dose of X842 once daily for five days based on safety and efficacy data generated from the previous cohort.
  Other Names: X842
  Arms: Multiple ascending dose of X842
Drug: Losec — Each subject in one cohort will be assigned to a standard dose of omeprazole once daily for five days.
  Other Names: omeprazole
  Arms: Losec

SUMMARY:
The purpose of this study is to assess and analyze the safety, tolerability and PK/PD data following single ascending and multiple ascending doses of X842 in healthy subjects.

DETAILED DESCRIPTION:
This is a single-centre, open label, first-in-human study with the primary objective to evaluate safety and tolerability of X842 after administration of single and multiple oral ascending doses to healthy male and female subjects. The study comprises a Single Ascending Dose (SAD) part and a Multiple Ascending Dose (MAD) part including an open-label multiple dose cohort administered active comparator (omeprazole). Four subjects will be included in each of the SAD and MAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study.
* Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 and weight at least 50 kg and no more than 100 kg at screening.
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
* Male subjects must be willing to use condom and if they have a fertile partner, she must use contraceptive methods with a failure rate of < 1% to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until three months after dosing of the IMP.
* Female subjects must be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal females defined as 12 months of amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulation hormone 25-140 IE/L and estradiol <200 pmol/L is confirmatory]).

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Present clinically significant psychiatric diagnosis, at discretion of the Investigator.
* Any clinically significant illness, medical/surgical procedure or trauma within four weeks of the first administration of investigational medical product.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years, regardless of whether there is evidence of local recurrence or metastases.
* History of any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs. The investigator is to be guided by evidence of any of the following: history of major gastrointestinal surgery such as gastrectomy, gastroenterostomy, bowel resection or Transjugular Intrahepatic Portosystemic Shunt (TIPS).
* History or presence of diagnosed and long-term treatment for GERD.
* Likelihood of having a gastric pH>2 due to for example known autoimmune gastritis or known Helicobacter pylori gastritis.
* Known severe atrophic gastritis.
* Vitamin B-12 deficiency and/or chronic Vitamin B-12 substitution.
* Known malabsorption.
* Any planned major surgery within the duration of the study.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
* After 10 minutes of supine rest at the time of screening, any vital signs values outside the following ranges:

  * Systolic BP 90 - 140 mm Hg
  * Diastolic BP 50 - 90 mm Hg
  * Heart rate (HR) 45-90 beats per minute
* Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
* History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to X842 or omeprazole.
* Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two weeks prior to the (first) administration of IMP, except occasional intake of paracetamol (maximum 2 000 mg/day; and not exceeding 6 000 mg/week), at the discretion of the Investigator and nasal decongestants without cortisone or antihistamine for a maximum of 10 days, at the discretion of the Investigator.
* Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment with less than three months between administration of last dose and first dose of IMP in this study. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
* Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
* Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP.
* Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse.
* Intake of xanthine and/or taurine containing energy drinks within two days prior to first day of IMP administration.
* Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Occurrence and frequency of AEs, changes in laboratory parameters, vital signs and physical examination after single and multiple doses of X842. Summary statistics will be applied. | Five weeks
  Safety and tolerability will be assessed by occurrence and frequency of AEs, changes in laboratory parameters, vital signs and physical examination. The adverse event assessment will follow the recommendations and grading system of Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Summary statistics will be applied.

SECONDARY OUTCOMES:
Measurement of the PK profile (Cmax) | Up to 48 hours after dosing
  To assess the Maximum Plasma Concentration (Cmax)
Measurement of the PK profile (t1/2) | Up to 48 hours after dosing
  To assess the plasma half life (t1/2) of drug
Measurement of the PD profile (intragastric pH) | Up to 24 hours after dosing
  To assess and characterize the PD profile with measurements of intragastric pH

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Lif-Tiberg, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- Clinical Trial Consultants, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson K, Carlsson E. Potassium-competitive acid blockade: a new therapeutic strategy in acid-related diseases. Pharmacol Ther. 2005 Dec;108(3):294-307. doi: 10.1016/j.pharmthera.2005.05.005. Epub 2005 Jul 5. PMID 16000224
- [Background] Hunt RH, Scarpignato C. Potassium-Competitive Acid Blockers (P-CABs): Are They Finally Ready for Prime Time in Acid-Related Disease? Clin Transl Gastroenterol. 2015 Oct 29;6(10):e119. doi: 10.1038/ctg.2015.39. PMID 26513137